CLINICAL TRIAL: NCT02094157
Title: An Open-Label Randomized Control Trial of Pre-Operative Low Molecular Weight Heparin Versus Tapered Warfarin as Bridging Therapy for Patients With Implantation of Pacemaker or Defibrillator
Brief Title: Tapered Warfarin or Interrupted Warfarin With Heparin Bridging for Pacemaker or Defibrillator Implantation
Acronym: PACEBRIDGE
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Change of practice made further recruitment impossible
Sponsor: McMaster University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PB 20080717
Record Dates: First submitted 2014-03-19; First posted 2014-03-21 (Estimated); Last update posted 2016-04-05 (Estimated); Status verified 2016-04

CONDITIONS: Cardiac Arrhythmias; Hemorrhage; Thromboembolism
Keywords: Atrial fibrillation; Mechanical heart valve; Stroke; Venous thromboembolism; Hemorrhage
MeSH Terms: conditions — Arrhythmias, Cardiac; Hemorrhage; Thromboembolism; Atrial Fibrillation; Stroke; Venous Thromboembolism | interventions — Heparin, Low-Molecular-Weight

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Bridged regimen (Active Comparator): Bridged regimen Warfarin therapy is stopped for 5 days before surgery and restarted in the evening of surgery at double the usual dose for two days. Bridging with low-molecular-weight heparin at therapeutic dose is given for 2½ days before surgery.
  Interventions: Drug: Bridged regimen Low-molecular-weight heparin
- Tapered warfarin regimen (Experimental): Tapered warfarin regimen Warfarin is given at half the usual maintenance dose for 3-6 days before surgery depending on the INR at the baseline visit. A double dose is given in the evening of surgery. No bridging with LMWH is used.
  Interventions: Drug: Tapered warfarin regimen

INTERVENTIONS:
Drug: Tapered warfarin regimen — This intervention is assigned to the experimental arm - Tapered warfarin regimen
  Other Names: Half dose warfarin
  Arms: Tapered warfarin regimen
Drug: Bridged regimen Low-molecular-weight heparin — This intervention is assigned to the active control arm - Bridged regimen
  Other Names: Low-molecular-weight heparin
  Arms: Bridged regimen

SUMMARY:
Approximately 2 million patients in North America are currently treated with the blood thinner warfarin. These patients have every year more than 200,000 invasive procedures, for which warfarin must be stopped to avoid bleeding complication. To protect the patient against blood clots and stroke while warfarin is stopped, most physicians today order "bridging" with low-molecular-weight heparin (LMWH). This is another blood thinner and it is injected under the skin during 3 days before the procedure. For implantation of pacemaker or defibrillator (27,000/year in Canada) the "bridging" routines vary a lot.The common "bridging" treatment with LMWH for 3 days before pacemaker surgery causes bleeding in the "pocket" where the pacemaker is placed in about 5%. For comparison, patients not on any blood thinners develop this bleeding in 2% after this surgery. "Pocket bleeding" may require evacuation of the blood collection and may cause infection. "Pocket bleeding" is thus a fairly common and clinically important but rarely a dangerous bleeding complication. It is a suitable safety endpoint in a study of "bridging" of blood thinners. LMWH costs $80-120, for which some patients are not covered. They have to be taught self-injection technique or have a nurse come to their home. The main hypothesis is if patients on blood thinners can be managed more conveniently before and after pacemaker surgery, without injections, without increased risk of pocket bleeding.

DETAILED DESCRIPTION:
Patients are recruited from those routinely referred before surgery for adjustment of their blood thinners. Suitable and consenting patients are randomized to one of the two regimens. They will either stop warfarin for 5 days and replace it with injections of LMWH for 3 days before pacemaker or implantable cardioverter defibrillator (ICD) surgery. The other group will have the dose of warfarin reduced to half for 3-6 days before surgery, depending on how thin their blood is. For all patients the degree of blood thinning is checked the day before surgery. If the blood is still to thin, the patient is instructed to take by mouth a dose of vitamin K, provided by us, to reduce the effect of warfarin. After surgery the patients restart warfarin at a double dose for 1 or 2 days to quickly reach the therapeutic effect again. Staff from the Pacemaker or Defibrillator Clinic, unaware of the treatment allocation, examines the patient for bleeding in the implantation pocket before they leave the hospital, and at routine follow-up after 2-3 weeks and 90 days.

ELIGIBILITY:
Inclusion Criteria:

* The patient has been receiving warfarin therapy for at least 1 week and is planned to continue this treatment for at least one month post-procedure
* The patient will have elective implantation or replacement of a pacemaker or ICD

Exclusion Criteria:

* Age <18 years
* Previous stroke
* Stroke risk (CHADS2) score of 0 or 1 in patients with atrial fibrillation as the only indication for anticoagulation
* Creatinine clearance (CrCl) <30 mL/min
* Surgery planned for a Monday or a day after a holiday
* Patient unsuitable for the study as assessed by the investigator (e.g., psychiatric disorder, history of non-compliance)
* Failure to obtain written consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 173 (Actual)
Dates: Start 2007-12; Primary Completion 2013-11 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
Pocket hematoma | 1 month
  Pocket hematoma is defined as palpable swelling of the pacemaker or defibrillator pocket exceeding the size of the generator.

SECONDARY OUTCOMES:
Major bleeding | 1 month
  Fatal bleeding OR Symptomatic bleeding in a critical area or organ, such as intracranial, intraspinal, intraocular, retroperitoneal, intraarticular or pericardial, or intramuscular with compartment syndrome OR Bleeding causing a fall in hemoglobin level of 20 g·L-1 (1.24 mmol·L-1) or more, or leading to transfusion of two or more units of whole blood or red cells.
Thromboembolism | 1 month
  Arterial thromboembolism, consisting of one or more of the following: stroke (ischemic or hemorrhagic), transient ischemic attack, systemic embolism to a limb or viscus, thrombosis of a mechanical or native heart valve, or thrombosis of a cardiac chamber. OR Venous thromboembolism that is symptomatic AND for deep vein thrombosis is verified by ultrasound, venography or computed tomography; for pulmonary embolism is verified by ventilation-perfusion lung scan, spiral computed tomography or pulmonary angiography.

OTHER OUTCOMES:
Preoperative reversal with vitamin K | 1 day
  Patients with International Normalized Ratio (INR) above 1.7 the day before surgery require correction of the coagulopathy with vitamin K to allow for surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Sam Schulman, MD, PhD, Principal Investigator — McMaster University
Locations (2):
- Canada (2):
  - Hamilton Health Sciences-General Hospital, Hamilton, Ontario
  - St. Joseph's Healthcare, Hamilton, Ontario

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Schulman S, Healey JS, Douketis JD, Delaney J, Morillo CA. Reduced-dose warfarin or interrupted warfarin with heparin bridging for pacemaker or defibrillator implantation: a randomized trial. Thromb Res. 2014 Oct;134(4):814-8. doi: 10.1016/j.thromres.2014.07.028. Epub 2014 Aug 1. PMID 25127655